CLINICAL TRIAL: NCT01434550
Title: Phase II Study of First-line Stereotactic Body Radiation Therapy (SBRT) in Patients With Non-Metastatic Unresectable Pancreatic Cancer
Brief Title: Phase II Study of First-line SBRT in Patients With Non-Metastatic Unresectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: research cancelled
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16459
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Tumor
Keywords: pancreas; pancreatic cancer; SBRT; stereotactic body radiation; radiation therapy; unresectable; non-metastatic; tissue, blood, research imaging; TBRI
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Histocompatibility Testing; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TBRI Subgroup: TBRI and SBRT (Active Comparator): Six patients will be asked to be part of a subgroup called TBRI (Tissue, Blood, Research Imaging). In this subgroup, we want to study if there is early death of tumor cells from the treatment by looking at the tumor using PET/CT scans and biopsies, and by testing the participant's body's white blood cells taken by a procedure called leukapheresis.
  Participants do not have to take part in the TBRI subgroup to get treatment on this study with SBRT.
  SBRT:
  1. 30 Gy in 5 fractions to pancreatic tumor
  2. 50 Gy in 5 daily consecutive fractions unresectable portion and avoiding bowel, stomach, and duodenum
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Radiation: Tissue, Blood, Research Imaging (TBRI)
- SBRT Alone (Active Comparator): 1. 30 Gy in 5 fractions to pancreatic tumor
  2. 50 Gy in 5 daily consecutive fractions unresectable portion and avoiding bowel, stomach, and duodenum
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Everyone who takes part in this study will receive SBRT. After making an individual radiation plan for each participant, they will receive 5 days of radiation to the pancreas. Participants will have follow-up visits with blood tests one month after the end of SBRT and then every 3 months for 3 years. They will also have CT scans (chest and pancreas) and FDG PET/CT (body) at 1 month and then at 3, 6, 9 and 12 months.
  Other Names: extracranial lesions; high-dose fractions; radiosurgery
Radiation: Tissue, Blood, Research Imaging (TBRI) — Post-SBRT procedures (day 1, 3, 5 of SBRT, and 4 weeks after) A) Endoscopic or CT guided biopsy of treated pancreatic cancer to assess
  1. Necrosis/apoptosis
  2. Lymphocyte infiltrate and antigen presenting cells B) Imaging to evaluate cell death (day 1, 3, 5 of SBRT, and 4 weeks after)
  1. Aposense-PET imaging
  Other Names: CT guided biopsy; Imaging to evaluate cell death; Aposense-PET imaging
  Arms: TBRI Subgroup: TBRI and SBRT

SUMMARY:
The purpose of this study is to see if SBRT will be a better way to treat pancreas cancer and to find out what effects, good and/or bad, this treatment will have on participants and their cancer.

DETAILED DESCRIPTION:
The standard treatment for cancer of the pancreas is surgery (if possible), external beam radiation therapy and/or chemotherapy. These standard treatments are not a cure and often extend life by just a few months. Recently, a new approach has been developed, called stereotactic body radiation therapy (SBRT). Based on the results of earlier studies using SBRT, the study doctors at Moffitt feel this is a reasonable alternative to the standard treatment for your disease.

Stereotactic body radiation therapy (SBRT) delivers high radiation doses to the tumor every day for 5 days which gives the usual 5-6 week course of radiation in less than a week. It has also been shown to have much less side effects.

The purpose of this study is to see if SBRT will be a better way to treat pancreas cancer and to find out what effects, good and/or bad, this treatment will have on you and your cancer.

Six patients will be asked to be part of a subgroup called TBRI (Tissue, Blood, Research Imaging). In this subgroup, the investigators want to study if there is early death of tumor cells from the treatment by looking at the tumor using PET/CT scans and biopsies, and by testing your body's white blood cells taken by a procedure called leukapheresis. You do not have to take part in the TBRI subgroup to get treatment on this study with SBRT.

ELIGIBILITY:
Inclusion Criteria - All Patients:

* Biopsy proven, non-metastatic, pancreatic cancer
* Unresectable disease based on institutional standardized criteria for unresectability
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* CT scan of chest and abdomen (3-phase pancreas protocol), and PET-CT within 4 weeks of study entry
* Patients with biliary or gastroduodenal obstruction must have drainage, duodenal stenting, or gastric bypass prior to initiating radiation
* All disease must be encompassed in a single radiation field
* No evidence or history of an autoimmune dysfunction
* Negative pregnancy test within 7 days of study entry
* No prior or concurrent chemotherapy
* No previous or concurrent immunotherapy for pancreatic cancer
* Liver enzymes ≤ 3 times upper limit of normal (ULN): total bilirubin (Tbili) ≤ 3.9 (biliary stents are allowed); aspartic transaminase (AST) ≤ 177; alanine transaminase (ALT) ≤ 198; Alkaline phosphatase (ALK-P) ≤ 378
* Adequate pretreatment organ function: Creatinine no greater than 1.5mg/dL; Total calcium no greater than 11.0mg/dL; prothrombin time (PT) no greater then 14 seconds; partial thromboplastin time (PTT) no greater then 40 seconds
* Ability to give informed consent
* Adequate baseline hematopoietic function: total white blood cell count equal to or greater than 3,000/mm³; absolute granulocyte count greater than 1,500/mm³; absolute lymphocyte count greater than 500/mm³; platelet count equal to or greater than 100,000/mm³

Inclusion Criteria - TBRI Group:

* All Participant inclusion criteria
* Amenable to leukapheresis as determined by a leukapheresis nurse
* Primary tumor that is accessible to direct intratumoral injection by CT-guidance confirmed by interventional radiologist
* No history of autoimmune disease
* No history of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS) or other immunosuppressive diseases
* No active viral or bacterial infection
* No use of steroids or any other immunosuppressive drug at least 4 weeks prior to enrollment on study

Exclusion Criteria - All Patients:

* Prior history of radiotherapy that overlaps with the planned ports to the primary pancreatic tumor
* Patients with tumors that are not accessible to direct access cannot be included in the study.
* Prior or concurrent chemotherapy
* Prior history of antineoplastic therapy or irradiation
* Prior treatment with anti-tumor vaccines not allowed
* Patients with a history of autoimmune diseases
* A history of HIV infection, AIDS or other immunosuppressive disease state. The need to exclude patients with HIV/AIDS is because one of the endpoints of the study is immune response. People with HIV have a compromised immune system and enrollment in this study could confound the results (TBRI only)
* Patients requiring corticosteroids are ineligible because one of the endpoints of the study is immune response. Since steroids modulate the immune system, enrollment of patients on steroids could confound the results. There must be no use of corticosteroids in the fours weeks preceding entry into the study (TBRI only).
* Active bacterial, fungal or viral infection
* Active bleeding (hemoptysis, melena, etc.)
* Women who are currently pregnant or actively breast feeding. Women of childbearing potential must have a negative serum pregnancy test and must use effective contraception during trial participation
* Any medical or psychiatric illness which in the opinion of the principal investigator might compromise a patient's ability to tolerate or complete treatment
* Any patient requiring blood thinners (due to risk of gastrointestinal [GI] bleed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Overall Survival (OS) | 36 Months
  Patients will be followed for 36 months to determine overall survival even after completion of the experimental portion of the protocol. Patients will be followed every 3 months. All patients will be referred for chemotherapy at the completion of radiation.

SECONDARY OUTCOMES:
Number of Participants With Reduction in Size of Primary Tumor | 12 Months
  Patients will undergo 64 slice helical computed tomography (CT) scan and feeding (FDG) pressure equalizing tube (PET)-CT scan pretreatment and at the conclusion of the study which will be separated by a 5 week time span. Subsequent helical CT and FDG PET-CT scans will be performed at 3, 6, 9 and 12 months with CA 19-9 levels. The Response Evaluation Criteria In Solid Tumors (RECIST) criteria will be used to measure clinical response. Time to local and distant disease progression will also be measured.
Number of Participants With Adverse Events (AEs) | 36 Months
  Toxicity response will be assessed and reported using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Shridhar, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute